CLINICAL TRIAL: NCT02092987
Title: Northern-Manhattan Hispanic Caregiver Intervention Effectiveness Study
Acronym: NHiCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Hebrew Home at Riverdale (Other); NYU Langone Health (Other); Burgio Geriatric Consulting (Unknown); Riverstone Senior Life Services (Unknown); Alzheimer's Association (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, José A. Luchsinger, Associate Professor of Medicine and Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AAAM5150; 7160 (Other: Patient-Centered outcomes Research Institute)
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2020-09

CONDITIONS: Depressive Symptoms; Burden
Keywords: Hispanic; Dementia; Caregivers; Depressive symptoms; Burden; Pragmatic randomized trial
MeSH Terms: conditions — Depression; Dementia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NYU Caregiver Intervention (Experimental): The New York University (NYU) caregiver intervention arm received the NYU caregiver intervention in addition to social work support and educational materials.
  Interventions: Other: Social work support; Other: Educational material; Behavioral: NYU caregiver counseling intervention
- REACH OUT (Active Comparator): The Resources for Enhancing Caregiver Health Offering Useful Treatments (REACH OUT) intervention arm received the REACH OUT caregiver intervention in addition to social work support and educational materials.
  Interventions: Other: Social work support; Other: Educational material; Behavioral: REACH OUT counseling intervention

INTERVENTIONS:
Other: Social work support — All study participants were provided access to social support services at Riverstone Senior Life services
Other: Educational material — All participants received educational material about dementia and caregiving in addition to information about resources for persons with dementia and their caregivers, including resources at the Alzheimer's Association such as support groups, and clinical and service resources available citywide.
Behavioral: NYU caregiver counseling intervention — The first component consists of 2 individual and 4 family counseling sessions. These sessions last between 1 and 1.5 hours. The second component of the intervention is participation in a caregiver support group . The third component of the treatment is "ad hoc" counseling. New psychiatric and behavioral problems of patients, which are generally more stressful than the need for assistance with activities of daily living or physical limitations, often precipitate ad hoc calls from caregivers.
  Arms: NYU Caregiver Intervention
Behavioral: REACH OUT counseling intervention — All aspects of the REACH OUT Intervention involve problem solving techniques and the development of written action plans. The goal of this intervention is to engage the caregiver in joint problem-solving with the objective of creating a written action plan targeting specific caregiving problems. The basic steps of problem solving are: 1.Define the problem. 2. Set goals 3. Brainstorm with caregiver and List possible solutions on a pad of paper, 4. Select solutions, 5. Develop an action plan based on these solutions, 6. Implement the action plan, track progress, and make adjustments as needed
  Arms: REACH OUT

SUMMARY:
The primary research question is which of the 2 best known dementia caregiver interventions, the New York University Caregiver intervention (NYUCI) and Resources for Enhancing Caregivers Health Offering Useful Treatments (REACH OUT), is more effective in alleviating depressive symptoms and caregiver burden among Hispanic caregivers in New York City. The investigators hypothesize that the NYUCI will be more effective than REACH OUT in reducing caregiver depressive symptoms and burden among Hispanics because of its focus on family-centered counseling, which is posited to be more important among Hispanic caregivers because of a cultural emphasis among Hispanics on family interactions in interventions. In order to answer the primary question, the investigators will conduct a pragmatic randomized trial comparing the NYUCI vs. REACH OUT in 200 Hispanic caregivers of persons with dementia in the community of Northern Manhattan. The total time of the intervention will be 6 months.

Our research question is which intervention, NYUCI or REACH OUT, is better in Hispanic relative (any relative) caregivers of persons with dementia. Our objective is to obtain effectiveness information that will help caregivers and health providers to make decisions about which intervention to choose. Our primary aim is to compare the effectiveness of the implementation of the NYUCI and REACH OUT in reducing depressive symptoms and burden. Our exploratory aims are to examine and compare the predictors of effectiveness of the NYUCI and REACH OUT and to examine additional outcomes such as caregiver stress and physical health, and outcomes related to the person with dementia. METHODS. We will conduct a pragmatic randomized trial of 200 relative caregivers of persons with dementia. Participants will be randomized to the NYUCI or REACH OUT. The total duration of the intervention will be 6 months, with assessments at baseline and follow-up. All interventions and questionnaires will be conducted in both English and Spanish. The study duration will be 3 years. The primary outcomes will be changes in caregiver depressive symptoms, measured with the Geriatric Depression Scale, and in caregiver burden using the Zarit caregiver burden interview.

DETAILED DESCRIPTION:
The prevalence of dementia is increasing with the aging of the population and the absence of prevention or cure. Thus, the burden of dementia on caregivers is also increasing. Hispanics have a higher prevalence of dementia than non-Hispanic Whites (NHW), have higher caregiving burden, and may have less economic resources to cope with the caregiving burden. However, there is a paucity of evidence on the effectiveness of caregiver interventions in Hispanics. We propose to compare 2 interventions with evidence of efficacy, the New York University Caregiver intervention (NYUCI) and the translated Resources for Enhancing Caregivers Health Offering Useful Treatments (REACH OUT). The NYUCI is a family centered counseling intervention that focuses on reducing negative family interactions and improving family support of the primary caregiver. REACH OUT focuses on caregiver skills training through action-oriented formal problem solving, goal setting, and written action plans. The effectiveness of the NYUCI and the REACH OUT has never been compared. Thus, there is no way for caregivers to decide which intervention to choose. In addition, there is a paucity of data on the effectiveness of both interventions in Hispanics.

ELIGIBILITY:
Inclusion Criteria:

* Self identified Hispanic
* Between the ages of 18 and 90.
* Caregiver is related to persons receiving care either as a spouse (including common law partners) or a blood or in-law relative.
* Person receiving care has been diagnosed with dementia and reports at least 1 memory/cognition and 1 daily functioning symptom in our screening questionnaire (see appendix).
* Caregiver is physically able to provide care
* Caregiver does not have a diagnosis of major psychiatric disorder other than depression.
* Caregiver does not have depression with psychotic features or suicidal ideation or attempts in the last 5 years.
* Caregiver is expected to live in New York City in the next 6 months or is available for study procedures in the New York City area.
* There is at least one relative or close friend living in the New York City Metropolitan Area (New York, New Jersey, Connecticut).

Exclusion Criteria:

* Not Hispanic
* Caregiver is not a relative as defined in the inclusion criteria.
* Person receiving care does not have dementia
* Other than depression, caregiver has a major psychiatric disorder such as schizophrenia
* Caregiver has depression with psychotic features or suicidal ideation in the last 5 years.
* Severe depression defined by a Patient Health Questionnaire (PHQ)-9 > 20.
* Previous or current participation in caregiver support programs with the NYUCI or the REACH OUT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Luchsinger, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luchsinger JA, Burgio L, Mittelman M, Dunner I, Levine JA, Kong J, Silver S, Ramirez M, Teresi JA. Northern Manhattan Hispanic Caregiver Intervention Effectiveness Study: protocol of a pragmatic randomised trial comparing the effectiveness of two established interventions for informal caregivers of persons with dementia. BMJ Open. 2016 Nov 25;6(11):e014082. doi: 10.1136/bmjopen-2016-014082. PMID 27888180

RESULTS

PARTICIPANT FLOW:
Groups:
- NYU Caregiver Intervention: The first component consists of 2 individual and 4 family counseling sessions. These sessions last between 1 and 1.5 hours. The second component of the intervention is participation in a caregiver support group . The third component of the treatment is "ad hoc" counseling. New psychiatric and behavioral problems of patients, which are generally more stressful than the need for assistance with activities of daily living or physical limitations, often precipitate ad hoc calls from caregivers.
  Social work support: All study participants will be provided access to social support services at Riverstone Senior Life services
  Educational material: All participants receive educational material about dementia and caregiving in addition to information about resources for persons with dementia and their caregivers, including resources at the Alzheimer's Association such as support groups, and clinical and service resources available citywide.
- REACH OUT: All aspects of the REACH OUT Intervention involve problem solving techniques and the development of written action plans. The goal of this intervention is to engage the caregiver in joint problem-solving with the objective of creating a written action plan targeting specific caregiving problems. The basic steps of problem solving are: 1.Define the problem. 2. Set goals 3. Brainstorm with caregiver and List possible solutions on a pad of paper, 4. Select solutions, 5. Develop an action plan based on these solutions, 6. Implement the action plan, track progress, and make adjustments as needed.
  Social work support: All study participants will be provided access to social support services at Riverstone Senior Life services Educational material: All participants receive educational material about dementia and caregiving in addition to information about resources for persons with dementia and their caregivers, including resources at the Alzheimer's Association such as support groups, a
Period: Overall Study
Arm/Group | NYU Caregiver Intervention | REACH OUT
Started | 110 | 111
Completed | 106 | 103
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NYU Caregiver Intervention | REACH OUT | Total
Number analyzed (Participants) | 110 | 111 | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.15 (11.28) | 58.33 (11.26) | 58.24 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 91 | 183
  Male | 18 | 20 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 110 | 111 | 221
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 110 | 111 | 221

OUTCOME MEASURES:

1. Primary Outcome: Score on Geriatric Depression Scale
Description: The Geriatric Depression Scale (GDS) is a 30-item self-report assessment used to identify depression in the elderly. The GDS questions are answered "yes" or "no", instead of a five-category response set. One point is assigned to each answer and the cumulative score is rated on a scoring grid. The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".Higher scores indicate more depressive symptoms.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYU Caregiver Intervention | REACH OUT
Number analyzed (Participants) | 110 | 111
units on a scale | 9.57 (7.12) | 9.80 (7.25)
Statistical Analysis 1: Comparison: NYU Caregiver Intervention vs REACH OUT; Hypothesis testing in changes in mean from baseline to follow-up were were conducted primarily with mixed models. Sensitivity analyses were conducted using ANOVA; Test type: Superiority or Other; p = 0.70, Mixed Models Analysis; interaction term

2. Primary Outcome: Score on Zarit Caregiver Burden Scale
Description: Zarit Caregiver Burden Scale measures caregiver burden by asking caregivers to respond to a series of 22 questions about the impact of the patient's disabilities on their life. For each item, caregivers are to indicate how often they felt that way (never, rarely, sometimes, quite frequently, or nearly always). The Burden Interview is scored by adding the numbered responses of the individual items. Higher scores indicate greater caregiver distress. Estimates of the degree of burden can be made from preliminary findings: 0 - 20 (little or no burden), 21 - 40 (mild to moderate burden), 41 - 60 (moderate to severe burden), and 61 - 88 (severe burden).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYU Caregiver Intervention | REACH OUT
Number analyzed (Participants) | 110 | 111
units on a scale | 36.24 (15.88) | 35.46 (18.04)
Statistical Analysis 1: Comparison: NYU Caregiver Intervention vs REACH OUT; Test type: Superiority or Other; p = 0.77, Mixed Models Analysis — comparison of arms using mixed models

3. Secondary Outcome: Score on Patient Reported Outcomes Measurement Information System (PROMIS) Physical Health Scale
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) Physical Health Scale: For adults, each question has five response options ranging in value from one to five (for pediatrics and parent proxy it is 0 to 4). To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 10-item form, the lowest possible raw score is 10; the highest possible raw score is 50. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A high score always represents more of the concept being measured. Higher scores indicate better health.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- NYU Caregiver Intervention: This arm received the NYU counseling intervention in addition to social work support and educational material
  Social work support: All study participants will be provided access to social support services at Riverstone Senior Life services
  Educational material: All participants receive educational material about dementia and caregiving in addition to information about resources for persons with dementia and their caregivers, including resources at the Alzheimer's Association such as support groups, and clinical and service resources available citywide.
- REACH OUT: This arm received the REACH OUT counseling intervention in addition to social work support and educational material
Arm/Group | NYU Caregiver Intervention | REACH OUT
Number analyzed (Participants) | 110 | 111
T-score | 30.10 (8.36) | 28.68 (7.38)
Statistical Analysis 1: Comparison: NYU Caregiver Intervention vs REACH OUT; Test type: Superiority or Other; p = 0.51, Mixed Models Analysis

4. Secondary Outcome: Score on Perceived Stress Scale (PSS)
Description: The Perceived Stress Scale is a self-report measure of stress that would be used to measure caregiver stress. The total score is calculated by finding the sum of 10 items, reverse coding questions 4, 5, 7, & 8. The PSS has a range of scores between 0 and 40. A higher score indicates more stress.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NYU Caregiver Intervention | REACH OUT
Number analyzed (Participants) | 110 | 111
units on a scale | 14.98 (8.10) | 14.95 (8.22)
Statistical Analysis 1: Comparison: NYU Caregiver Intervention vs REACH OUT; Test type: Superiority or Other; p = 0.51, Mixed Models Analysis

5. Secondary Outcome: Score on the PROMIS Short Form (SF) Depression Scale
Description: Depressive symptoms measured with the PROMIS SF Depression Scale: Each question has five response options ranging in value from one to five. To find the total raw score, sum the values of the response to each question. For example, for the eight-item form, the lowest possible raw score is 8; the highest possible raw score is 40. The total raw score is then converted into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher score means more depressive symptoms.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | NYU Caregiver Intervention | REACH OUT
Number analyzed (Participants) | 110 | 111
T-score | 48.01 (10.32) | 48.51 (10.28)
Statistical Analysis 1: Comparison: NYU Caregiver Intervention vs REACH OUT; Test type: Superiority or Other; p = 0.76, Mixed Models Analysis

6. Secondary Outcome: Total Score on Patient Health Questionnaire (PHQ-9)
Description: The PHQ-9 is the depression module, which scores each of the 9 Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria as "0" (not at all) to "3" (nearly every day). PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively. The range of the total score of the PHQ-9 is 0 to 27, with higher scores indicating more depressive symptoms.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NYU Caregiver Intervention | REACH OUT
Number analyzed (Participants) | 110 | 111
score on a scale | 5.40 (5.40) | 4.73 (4.49)
Statistical Analysis 1: Comparison: NYU Caregiver Intervention vs REACH OUT; Test type: Superiority or Other; p = 0.79, Mixed Models Analysis

7. Other Pre Specified Outcome: Score on the Lawton Caregiving Appraisal Scale (CAS) - Burden Subscale
Description: The Lawton Caregiver Appraisal Scale burden subscale has 9 items. Items include "Do you feel that because of the time you spend with your Elder that you don't have enough time for yourself?", "Do you feel your health has suffered because of your involvement with your Elder?," "Do you feel that your social life has suffered because you are caring for your Elder?", "Do you feel that you will be unable to take care of your Elder much longer?", "Do you feel you have lost control of your life since your Elder's illness?", "Do you feel very tired as a result of caring for your Elder?", "Do you feel isolated and alone as a result of caring for your Elder?", "Taking care of my Elder gives me a trapped feeling", and "I can fit in most of the things I need to do in spite of the time taken by caring for my Elder". The five-point Likert scale responses ranged from "never" to "nearly always." The score ranges from 5 to 45; higher score indicates greater burden
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NYU Caregiver Intervention | REACH OUT
Number analyzed (Participants) | 110 | 111
score on a scale | 23.42 (8.72) | 23.73 (9.26)
Statistical Analysis 1: Comparison: NYU Caregiver Intervention vs REACH OUT; Test type: Superiority or Other; p = 0.62, Mixed Models Analysis

8. Other Pre Specified Outcome: Score on Montgomery Objective Burden Scale
Description: The Montgomery Caregiving Objective Burden Scale consists of 6 items. Caregivers are asked if caregiving responsibilities have "decreased time you have to yourself", "given you little time for friends and relatives", "caused your social like to suffer", "changed your routine", "left you with almost no time to relax", and "kept you from recreational activities". Items were rated on a five point Likert scale ranging from "not at all" to "a great deal". The score ranges from 5 to 30; Higher score indicates greater burden
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NYU Caregiver Intervention | REACH OUT
Number analyzed (Participants) | 110 | 111
score on a scale | 18.00 (7.10) | 17.26 (6.84)

ADVERSE EVENTS:
Arm/Group | NYU Caregiver Intervention | REACH OUT
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/111
Other Adverse Events (participants affected / at risk) | 0/110 | 0/111

LIMITATIONS AND CAVEATS:
The study was designed with a relatively short follow-up of 6 months which may have been too short to observe any significant chance in depressive symptoms. In addition, anxiety was not measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No